CLINICAL TRIAL: NCT05979181
Title: Peripartum Cesarean Hysterectomy for Placenta Percreta: a Retrospective Analysis of Cases With and Without Extrauterine Disease
Brief Title: Peripartum Cesarean Hysterectomy for Placenta Percreta
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: R.23.06.2211
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Placenta Accreta
Keywords: PAS; Placenta previa; Placenta accreta; Cesarean hysterectomy
MeSH Terms: conditions — Placenta Accreta; Placenta Previa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No extrauterine disease group: Women having placenta previa percreta with no extrauterine disease (FIGO grade 3a)
  Interventions: Procedure: Cesarean hysterectomy
- Extrauterine disease group: Women having placenta previa percreta with extrauterine disease (FIGO grades 3b and 3c)
  Interventions: Procedure: Cesarean hysterectomy

INTERVENTIONS:
Procedure: Cesarean hysterectomy — Cesarean hysterectomy due to placenta previa percreta with no extrauterine disease (FIGO grade 3a) or with extrauterine disease (FIGO grades 3b and 3c)

SUMMARY:
The aim of this study is to address the possible preoperative determinants of extrauterine diseases in cases of placenta previa percreta and to compare the operative and postoperative characteristics of cases with and without extrauterine disease.

DETAILED DESCRIPTION:
This will be a retrospective study of the data of women who underwent cesarean hysterectomy on placenta previa percreta who were classified as Federation of Gynecology and Obstetrics (FIGO) grade 3. Women without extrauterine disease (FIGO grade 3a) will be compared to women with extrauterine disease (FIGO grades 3b and 3c)

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent cesarean hysterectomy on placenta previa percreta (FIGO grade 3).

Exclusion Criteria:

* Medical conditions complicating pregnancy.
* Blood diseases or bleeding tendencies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who underwent cesarean hysterectomy on placenta previa percreta (FIGO grade 3) diagnosed by color flow Doppler, and confirmed intraoperatively
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Estimated amount of intraoperative blood loss | From start to end of operation
  Calculated amount of blood loss during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Khaled S Ismail, MD, Principal Investigator — Mansoura University; Mahmoud M Awad, MD, Study Director — Mansoura University; Alhussein A Mohamed, MD, Study Director — Mansoura University; Mohamed S Abdelhafez, MD, Study Chair — Mansoura University
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt